CLINICAL TRIAL: NCT01482637
Title: Improving Ethics in Research: Development of the Coercion Assessment Scale
Brief Title: Development of Coercion Assessment Scale
Acronym: CAS
Status: Completed | Type: Observational
Sponsor: Treatment Research Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: Public Health Management Corporation (Other)
Other Study IDs: #0902; R01DA025687 (NIH)
Record Dates: First submitted 2011-11-28; First posted 2011-11-30 (Estimated); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Coercion to Participate in Research

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- CAS: There are no separate groups. All subjects are being asked to complete the CAS measure.
  Interventions: Other: CAS

INTERVENTIONS:
Other: CAS — All clients will be asked to complete the CAS instrument.

SUMMARY:
In this study, the investigators seek to further develop the CAS as a comprehensive, reliable, and valid instrument for measuring coercion to participate in research among adult substance abusing offender populations.

DETAILED DESCRIPTION:
First, the investigators wish to widen the scope of the CAS so that it can reliably and validly measure perceived coercion. The content domain will be expanded to included pressures experienced by a range of individuals involved in the criminal justice system. Second, the investigators will finalize the CAS by ensuring that the instrument is appropriate for use with substance abusing offenders. A final goal of the study examines the psychometric properties of the instrument. This evaluation will include an examination of test-retest reliability, internal consistency and factor structure, and convergent and discriminant validity.

This study will be carried out in three distinct phases to satisfy the goals detailed above. The purpose of Phase 1 is to add to the already existing content of the CAS. In this phase, focus groups will be conducted with clients (i.e., substance abusing offenders) and professionals (i.e., treatment and criminal justice staff and stakeholders) in several different criminal justice. The goal of these groups will be to identify additional sources of coercion that substance abusing offenders may experience related to participation in research. The purpose of Phase 2 is to finalize and ensure the appropriateness of the instrument. In this phase, the investigators will conduct a protocol analysis with 30 drug court clients. The interviewer will read each item aloud to participants, and participants will provide their response. After completing each item, they will be interviewed about how they arrived at their decision. The purpose of Phase 3 is to evaluate the psychometric properties of the CAS. A total of 200 substance abusing offenders participating in an ongoing NIDA-funded study (i.e., the "host study") will receive TRI's manualized written informed consent procedure as part of their participation in the host study. Following consent, research staff will administer study assessments to all consented participants. Additionally, a random sample of 50 clients will be selected to complete a retest interview, scheduled three to five days following the initial interview to assess the extent to which responses vary between the two administrations.

ELIGIBILITY:
Inclusion Criteria:

* Virtually any defendant admitted to either the misdemeanor drug court of the New Castle County Court of Common Pleas, the 17th Judicial District Drug Court in Union and Snyder Counties, or any research participant in the NITE Study at Miriam Hospital will be eligible to participate.
* The legal criteria for entry into drug court require defendant to (1) be 18 years of age or older; (2)be a resident of or commit their offense in either New Castle County, Delaware or Union and Snyder Counties, respectively; (3) be charged with a misdemeanor drug offense including possession or consumption of cannabis, possession of drug paraphernalia, possession of hypodermic syringes, or driving under the influence (DUI); and (4) not have a history of a violent offense involving serious injury to a victim or use of a deadly weapon. Individuals with medical or psychiatric conditions will be eligible to participate in the study so long a they are capable of giving competent, informed consent to research participation.

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: For Phase 3, a total of 228 clients were drawn from the host study recruiting from a misdemeanor drug court in New Castle County, Delaware and from Miriam Prison in Rhode Island. The sample is representative of the combined demographic characteristics of our host studies with the study participants being 75% male, 75% Caucasian, and 22% African-American in the Wilmington and Rhode Island sites. Our sample of adolescents is representative of the host study with 78% African-American, 8% Caucasian and 13% "Other."
Sampling Method: Probability Sample
Enrollment: 228 (Actual)
Dates: Start 2010-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Expand Scope of CAS Measure | Months 9-30
  To expand the scope of the CAS so that it can reliably and validly measure perceived coercion to enter research studies in a wide-range of substance abusing offender populations. The content domain will be expanded to include pressures experienced by individuals who have been arrested but not adjudicated (i.e., drug court clients), offenders who have been adjudicated but are not currently incarcerated (i.e., parolees/probationers) and offenders who are currently incarcerated.
Ensuring CAS Use with Substance Abusing Offenders | Months 9-30
  To finalize the development of the CAS by ensuring that the instrument is appropriate for use with substance abusing offenders. Items on the instrument will be evaluated to ensure that they are correctly worded and that their intended meaning is accurately conveyed to participants.
Evaluate Psychometric Properties of CAS | Months 9-30
  To evaluate the psychometric properties of the CAS to ensure that it is a reliable and valid measure of perceived coercion to participate in research. The psychometric evaluation will include an examination of test-retest reliability, internal consistency and factor structure, and convergent and discriminant validity.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Dugosh, Ph.D., Principal Investigator — Treatment Research Institute
Locations (1):
- Treatment Research Institute, Philadelphia, Pennsylvania, United States